CLINICAL TRIAL: NCT00637169
Title: Efficacy and Safety of Targeting Lower Arterial Oxygen Saturations to Reduce Oxygen Toxicity and Oxidative Stress in Very Preterm Infants: The Canadian Oxygen Trial (COT)
Brief Title: Canadian Oxygen Trial (COT)
Acronym: COT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTG-2006-COT; MCT-79217/ISRCTN62491227
Record Dates: First submitted 2008-03-06; First posted 2008-03-17 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2014-12

CONDITIONS: Respiratory Insufficiency of Prematurity
Keywords: oxygen therapy; neurodevelopmental impairment
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Supplemental oxygen to maintain functional arterial oxygen saturations in the range of 85-89%. Dose of oxygen is determined by the individual infant's need to achieve the target oxygen saturations.
  Interventions: Other: Titration of oxygen therapy
- 2 (Active Comparator): Supplemental oxygen to maintain functional arterial oxygen saturations in the range of 91-95%. Dose of oxygen is determined by the individual infant's need to achieve the target oxygen saturations.
  Interventions: Other: Titration of oxygen therapy

INTERVENTIONS:
Other: Titration of oxygen therapy — Supplemental oxygen to maintain functional arterial oxygen saturations in one of two saturation target ranges.
  Other Names: Masimo Radical Pulse Oximeter

SUMMARY:
Study Question: In infants who are born at gestational ages of 23 0/7 to 27 6/7 weeks, does lowering the concentration of supplemental oxygen to target an arterial oxygen saturation by pulse oximetry (SpO2)of 85-89% compared with 91-95%, from the day of birth until the baby's first discharge home, increase the probability of survival without severe neurosensory disability to a corrected age of 18 months?

DETAILED DESCRIPTION:
Most extremely preterm babies require supplemental oxygen for several weeks or even months after birth. The goal of oxygen therapy is to achieve adequate oxygen delivery to the tissues without causing oxygen toxicity and oxidative stress. At present, this goal is elusive in very immature infants. Although it is standard practice in modern neonatal intensive care units to monitor arterial oxygen saturations via pulse oximetry, there is insufficient evidence to guide the choice of the upper and lower alarm limits. A rigorous trial with long-term follow up is urgently needed and long overdue to determine whether oxygen exposure can be reduced safely in extremely preterm infants without increasing the risk of hypoxic death or disability.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 23 0/7 - 27 6/7 weeks
* Postnatal age < 24 hours

Exclusion Criteria:

* Infant not considered viable (decision made not to administer effective therapies)
* Dysmorphic features or congenital malformations that adversely affect life expectancy or neurodevelopment
* Known or strongly suspected cyanotic heart disease
* Persistent pulmonary hypertension, e.g. associated with pulmonary hypoplasia
* Unlikely to be available for long-term follow-up

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1201 (Actual)
Dates: Start 2006-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survival without severe neurosensory disability to 18 to 21 months (corrected for prematurity) | 18-21 months corrected for prematurity

SECONDARY OUTCOMES:
Retinopathy of prematurity | 32 to 44 weeks postmenstrual age
Bronchopulmonary dysplasia | 36 weeks postmenstrual age
Brain injury | from week one of life up to 36 weeks postmenstrual age
Patent ductus arteriosus | until first discharge home
Necrotizing enterocolitis | until first discharge home
Growth | until 18-21 months corrected for prematurity
respiratory morbidity | until 18-21 months corrected for prematurity
Mean developmental index scores on the Bayley Scales | 18-21 months corrected for prematurity

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Schmidt, MD, Study Chair — McMaster University; Robin Roberts, MMath, Principal Investigator — Hamilton Health Sciences/McMaster University; Elizabeth Asztalos, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Alfonso Solimano, MD, Principal Investigator — Children's & Women's Health Centre of BC; Robin Whyte, MD, Principal Investigator — IWK Health Centre; Jack Rabi, MD, Principal Investigator — Foothills Hospital; Christian Poets, MD, Principal Investigator — University Children's Hospital Tuebingen
Locations (23):
- United States (3):
  - Stony Brook University Medical Center, Stony Brook, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania (HUP), Philadelphia, Pennsylvania
- Hospital Sanatorio de la Trinidad & Buenos Aires NICU Network, Buenos Aires, Argentina
- Canada (14):
  - Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - B.C. Children's Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario and Ottawa General Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - CHU Ste. Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Oulu University Central Hospital, Oulu, Finland
- University Children's Hospital, Tübingen, Germany
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Bnai-Zion Medical Center, Haifa
  - Meir Medical Center, Kfar Saba

REFERENCES:
- [Result] Schmidt B, Whyte RK, Asztalos EV, Moddemann D, Poets C, Rabi Y, Solimano A, Roberts RS; Canadian Oxygen Trial (COT) Group. Effects of targeting higher vs lower arterial oxygen saturations on death or disability in extremely preterm infants: a randomized clinical trial. JAMA. 2013 May 22;309(20):2111-20. doi: 10.1001/jama.2013.5555. PMID 23644995
- [Result] Schmidt B, Roberts RS, Whyte RK, Asztalos EV, Poets C, Rabi Y, Solimano A, Nelson H; Canadian Oxygen Trial Group. Impact of study oximeter masking algorithm on titration of oxygen therapy in the Canadian oxygen trial. J Pediatr. 2014 Oct;165(4):666-71.e2. doi: 10.1016/j.jpeds.2014.05.028. Epub 2014 Jun 25. PMID 24973289
- [Derived] Jensen EA, Whyte RK, Schmidt B, Bassler D, Vain NE, Roberts RS; Canadian Oxygen Trial Investigators. Association between Intermittent Hypoxemia and Severe Bronchopulmonary Dysplasia in Preterm Infants. Am J Respir Crit Care Med. 2021 Nov 15;204(10):1192-1199. doi: 10.1164/rccm.202105-1150OC. PMID 34428130